CLINICAL TRIAL: NCT03531502
Title: Initial Management of Patients Receiving a Single Shock (IMPRESS)
Acronym: IMPRESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Saint Luke's Health System (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPRESS
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Ventricular Tachycardia
Keywords: tachycardia; defibrillator; arrythmia
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard medical therapy (Active Comparator): Patients who have a positive NIPS study and are randomized to the medical therapy arm will either be initiated on antiarrhythmic therapy or will have their antiarrhythmic therapy intensified. All medication therapy is considered usual standard therapy.
  Interventions: Other: Standard Medical Therapy; Procedure: Non-Invasive Programmed Stimulation (NIPS)
- Ventricular Tachycardia Ablation (Experimental): Patients who have a positive NIPS study and are randomized to the ablation arm will undergo ventricular tachycardia ablation procedure guided by CardioInsight.
  Interventions: Procedure: Ventricular Tachycardia Ablation; Procedure: Non-Invasive Programmed Stimulation (NIPS)
- Negative NIPS/Non-intervention (Other): Patients who had a negative NIPS study will not be assigned to a treatment group and will be followed according to standard of care.
  Interventions: Procedure: Non-Invasive Programmed Stimulation (NIPS)

INTERVENTIONS:
Procedure: Ventricular Tachycardia Ablation — Ventricular Tachycardia Ablation
  Arms: Ventricular Tachycardia Ablation
Other: Standard Medical Therapy — For the antiarrhythmic naïve patients, the attending physician may initiate therapy with sotalol or amiodarone. For patients already on therapy with sotalol or amiodarone, the attending physician may choose to either increase the dosage/ frequency of these medications and/or add mexiletine to the regimen. Other alterations to medical therapy, such as adjusting the dose of beta-blockers, calcium-channel blockers, anti-hypertensive, diuretic or anti-anginal medications may be performed at the discretion of the attending physician.
  Arms: Standard medical therapy
Procedure: Non-Invasive Programmed Stimulation (NIPS) — All patients will receive this procedure in attempt to induce ventricular tachycardia. The outcome of this procedure determines if a patient will be randomized.

SUMMARY:
The goal of this study is to determine the optimal treatment for patients who receive a single shock from their implantable cardioverter defibrillator (ICD). All participants in this study will be fitted with a special electrode vest to detect the origin of heart rhythm abnormalities and then they will undergo a procedure called Non-Invasive Programmed Stimulation (NIPS). This procedure involves sedating a participants with anesthesia and then using the participant's own ICD to try to stimulate the heart to go into ventricular tachycardia. If this procedure is unable to induce the participant into ventricular tachycardia, then the participant will just be managed with usual care and will not be placed on any additional medications and will not undergo an ablation. However, if the NIPS induces the ventricular tachycardia, the electrode vest will be used to determine the origin of the abnormal heart rhythm inside the heart. After a successful NIPS procedure, the participants will be randomly assigned to either be placed on medication therapy or undergo catheter ablation. The outcomes from all three groups will be compared and the researchers hope to better understand which participants are most likely to benefit from watchful waiting versus medication versus catheter ablation.

DETAILED DESCRIPTION:
Patients with a history of ventricular tachycardia requiring defibrillation or who are at risk for developing ventricular tachycardia will undergo placement of an implantable cardioverter defibrillator (ICD) for purposes of prevention of sudden cardiac arrest. While the ICD is lifesaving, if a patient receives a shock from their ICD it is painful and the entire experience is very traumatic. Traditionally, the management of these patients who receive a single shock from their ICD is variable because it is not known if the patient will continue to experience further shocks or not. Some physicians will initiate antiarrhythmic medical therapy after only a single shock, whereas others will wait until the patient has recurrent ICD shocks before initiating therapy. All patients should be counseled to not drive for 6 months following a shock. Ventricular tachycardia ablation, a procedure involving placing catheters from the groin into the chambers of the heart to isolate the source of ventricular tachycardia and eliminate these foci through delivery of radiofrequency energy, is typically reserved for patients with multiple recurrent cases of ventricular tachycardia. While some studies have shown that ventricular tachycardia ablations can be done safely at an earlier course of the disease and this procedure has been demonstrated to reduce further ICD shocks, this practice is not commonplace.

Patients who undergo a ventricular tachycardia ablation procedure, will initially have catheters placed into the ventricular chambers of the heart and these catheters will be used to stimulate the heart in an attempt to induce the ventricular tachycardia, a process known as programmed stimulation. One major limitation of a ventricular tachycardia ablation procedure is the need to be able to induce the ventricular tachycardia rhythm via programmed stimulation. If this rhythm cannot be induced then it is very difficult to perform the ventricular tachycardia ablation procedure. Non-invasive programmed stimulation (NIPS) is a means of performing programmed stimulation using the patient's own ICD and does not involve placing catheters into the heart.

Aim: The aim of this study is to investigate if non-invasive programmed stimulation (NIPS) can be used to risk stratify patients determine if earlier intervention with either antiarrhythmic medications or ablation in patients with recurrent ventricular tachycardia that received ICD shocks would help decrease further ICD shocks and hospitalizations for ventricular arrhythmias.

Primary hypothesis: Patients receiving a single ICD shock for ventricular tachycardia who undergo a non-invasive programmed stimulation (NIPS) that fails to induce any sustained ventricular tachycardia, are at low likelihood of experiencing recurrent ICD shocks within the next year.

Secondary hypothesis: For patients receiving a single ICD shock for ventricular tachycardia who undergo non-invasive programmed stimulation (NIPS) that induces a sustained, monomorphic ventricular tachycardia rhythm, the performance of ventricular tachycardia ablation will reduce the incidence of recurrent ICD shocks within the next year, as compared to antiarrhythmic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old, both males and females
* Single or dual chamber ICD or BiVentricular ICD in situ
* Ischemic or non-ischemic cardiomyopathy
* Receive a single shock from their ICD for monomorphic ventricular tachycardia

Exclusion Criteria:

* ICD shock for polymorphic VT/VF or inappropriate shock
* Previous ventricular tachycardia ablation within 1 year
* NYHA Class IV heart failure or current inotrope therapy
* Ventricular tachycardia storm
* Listed for heart transplant or LVAD
* Pregnant as determined by urine pregnancy test prior to NIPS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
ICD Shocks | 12 months
  Number of recurrent ICD shocks

SECONDARY OUTCOMES:
Total Mortality | 12 months
  Number of related deaths
Hospitalizations | 12 months
  Number of related hospitalizations
ATP Therapy as recorded by ICD | 12 months
  Number of ATP therapies administered by ICD
Non-sustained VT | 12 months
Initiation of antiarrythmic medication | 12 months
  Number of times new medical therapy was started as documented in the medical record
Modification of antiarrythmic medication | 12 months
  Number of times medical therapy was changed
Repeat ablation | 12 months
  Number of repeat ablation procedures

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya Gupta, MD, Principal Investigator — Saint Luke's Health System
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Result] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Result] Frankel DS, Mountantonakis SE, Zado ES, Anter E, Bala R, Cooper JM, Deo R, Dixit S, Epstein AE, Garcia FC, Gerstenfeld EP, Hutchinson MD, Lin D, Patel VV, Riley MP, Robinson MR, Tzou WS, Verdino RJ, Callans DJ, Marchlinski FE. Noninvasive programmed ventricular stimulation early after ventricular tachycardia ablation to predict risk of late recurrence. J Am Coll Cardiol. 2012 Apr 24;59(17):1529-35. doi: 10.1016/j.jacc.2012.01.026. PMID 22516442
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933